CLINICAL TRIAL: NCT07338201
Title: The Effect of Video-Technology-Based Structured Self-Assessment on Nursing Students' Knowledge, Skills, and Self-Confidence in Peripheral Intravenous Catheter (PIVC) Insertion
Brief Title: The Effect of Video-Supported Self-Assessment on Nursing Students' Knowledge, Skills, and Self-Confidence in PIVC Insertion
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alev Keskin (Other)
Collaborators: Cukurova University (Other)
Responsible Party: Sponsor-Investigator, Alev Keskin, Sponsor-Investigator, Cukurova University
Organization: Cukurova University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: CU-PIVC-2025
Record Dates: First submitted 2025-11-18; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Clinical Skill Training - Peripheral IV Catheter Insertion
Keywords: Peripheral intravenous catheter; PIVC training; Nursing students; Video-assisted education; Structured self-assessment

STUDY DESIGN:
Intervention Model Description: Participants will be randomized into two parallel groups: intervention and control
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Students will receive video-assisted structured self-evaluation. Their PIVC insertion procedures will be video-recorded by the research team, reviewed by the students, followed by completion of a structured self-evaluation checklist and a guided feedback session.
  Interventions: Behavioral: Video-Assisted Structured Self-Evaluation
- Control Group (Active Comparator): Students will receive standard theoretical and practical PIVC training. Their procedures will also be video-recorded by the research team for assessment; however, students will not have access to their videos and will not perform structured self-evaluation.
  Interventions: Other: Standard Training

INTERVENTIONS:
Behavioral: Video-Assisted Structured Self-Evaluation — A behavioral educational method combining video-recorded performance review, structured self-evaluation, and guided feedback to improve PIVC knowledge, skills, and self-confidence.
  Arms: Intervention Group
Other: Standard Training — Participants receive standard theoretical and practical PIVC training without access to video review or structured self-evaluation.
  Arms: Control Group

SUMMARY:
This study aims to examine the effect of combining video-recorded performance with structured self-evaluation on nursing students' knowledge, skills, and self-confidence related to peripheral intravenous catheter (PIVC) insertion. In the intervention group, students' PIVC insertion procedures will be recorded by the research team. Students will watch their own performance videos, complete a structured self-evaluation checklist, and then participate in a guided feedback session. In the control group, students' procedures will also be video-recorded by the research team; however, they will not have access to their videos and will not perform self-evaluation. Outcomes will be assessed at baseline, immediately after the intervention, and at a two-week follow-up.

DETAILED DESCRIPTION:
Peripheral intravenous catheter (PIVC) insertion is a fundamental psychomotor skill in nursing education, yet students often experience anxiety, low confidence, and difficulty achieving competency during this learning process. Video-assisted structured self-evaluation is a contemporary educational method that enables students to review their own performance, increase self-awareness, identify errors, and refine their clinical decision-making.

This randomized controlled, parallel-group, assessor-blinded study investigates the impact of video-based structured self-evaluation on first-year nursing students' knowledge, technical skills, and self-confidence in PIVC insertion. In the intervention group, students' PIVC insertion performances during the skills laboratory session will be recorded by the research team. Students will then review their individual performance videos, complete a standardized structured self-evaluation checklist, and receive a guided feedback session from the instructor.

In the control group, students' PIVC insertion procedures will similarly be video-recorded by the research team for assessment purposes; however, students will not access their videos and will not complete structured self-evaluation or receive video-based feedback.

Knowledge levels, skill performance, and self-confidence will be measured at three time points: baseline (pretest), immediately after the training session (posttest), and two weeks later (follow-up). Skill performance scores will be obtained through blinded evaluation of the video recordings using a standardized PIVC skills checklist.

ELIGIBILITY:
Inclusion Criteria:

* Being a first-year nursing student

  * Learning and performing peripheral intravenous catheter (PIVC) insertion for the first time
  * Voluntarily agreeing to participate in the studyo

Exclusion Criteria:

* Being a 2nd-, 3rd-, or 4th-year nursing student

  * Having prior knowledge of peripheral intravenous catheter (PIVC) insertion or having previously performed the procedure
  * Failure to comply with the study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
PIVC Knowledge Score | Baseline (Day 0, prior to training), immediately post-training (Day 1) and 2 weeks after training
  A 20-item multiple-choice theoretical knowledge test developed by the researchers to assess students' knowledge of peripheral intravenous catheter (PIVC) insertion. Scores range from 0 to 100, with higher scores indicating greater PIVC knowledge.
PIVC Skill Performance Score | immediately post-training (Day 1) and 2 weeks after training
  A 47 item PIVC skill checklist developed based on CDC guidelines and expert review, assessing students' practical performance during PIVC insertion. Each item is scored as 1 (performed correctly) or 0 (not performed), with total scores ranging from 0 to 47 Higher scores indicate better PIVC skill performance
PIVC Self-Confidence Score | Baseline (Day 0, prior to training), immediately post-training (Day 1) and 2 weeks after training
  The 15-item Peripheral Intravenous Catheter Insertion Self-Confidence Scale (Marchionni et al., 2024; Turkish validity by Özbay et al., 2025) assessing students' confidence in learning and performing PIVC insertion. Items are rated on a 5-point Likert scale (1-5), with higher scores indicating higher self-confidence.

OTHER OUTCOMES:
Demographic Information Form | Baseline (Day 0, prior to training)

IPD SHARING:
Plan to Share IPD: No